CLINICAL TRIAL: NCT04039152
Title: Clinical Impact of an Antibiotic Stewardship Program in a Neonatal Intensive Care Unit at a Tertiary Care Hospital: A Prospective Quasi Experimental Clinical Study
Brief Title: Clinical Impact of an Antibiotic Stewardship Program in a Neonatal Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Neveen Hassan, Principle investigator, Assiut University
Other Study IDs: AssiutUU
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Neonatal Sepsis
Keywords: Antibiotics; Antimicrobial resistance; Antibiotic stewardship program; Neonatal intensive care unit; Neonatal sepsis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The pre-antibiotics stewardship program phase: This phase included making NICU-specific antibiograms, choosing the antibiotic use evaluation measures, conducting antibiotic use evaluations, and designing the antibiotics stewardship program (ASP).
- The antibiotics stewardship program intervention phase: The ASP intervention phase included implementation of the ASP, which involved modifying the neonatal sepsis treatment protocol according to the local antibiotic susceptibility patterns and measuring its clinical outcomes.
  Interventions: Other: locally adapted neonatal sepsis treatment protocol

INTERVENTIONS:
Other: locally adapted neonatal sepsis treatment protocol — the neonatal sepsis treatment protocol was modified according to the local antibiotics susceptibility patterns
  Other Names: implementing a new antibiotic dosing protocol, increasing the number of ordered microbiological cultures, the number of C-reactive protein (CRP) tests per patient.
  Groups: The antibiotics stewardship program intervention phase

SUMMARY:
Antimicrobial resistance is one of the biggest and most urgent threat to global health. Initiating antimicrobial stewardship programs is one of the main efforts to control antimicrobial resistance. Implementing these programs in neonatal intensive care units (NICU)is very important and crucial despite of its difficulty, where antibiotics are used extensively. The aim of present study was to assess the clinical impact of implementing antibiotic stewardship program interventions at NICU.

DETAILED DESCRIPTION:
Background:

Implementing an antimicrobial stewardship program is one of the main efforts to control antimicrobial resistance. The present study aimed to assess the clinical impact of the antibiotics stewardship program (ASP) in the neonatal intensive care unit (NICU) of Assiut University Children's Hospital.

Methods:

The study was conducted in two phases from January 2019 to June 2020. The pre-ASP phase (603 patients) included making NICU-specific antibiograms, choosing the antibiotic use evaluation measures, conducting antibiotic use evaluations, and designing the ASP. The ASP intervention phase (597 patients) included implementation of the ASP, which involved modifying the neonatal sepsis treatment protocol according to the local antibiotic susceptibility patterns and measuring its clinical outcomes.

Results:

The ASP intervention phase showed a significant increase in the number of C-reactive protein tests, microbiological cultures/patient, the number of patients taking definitive therapy, and the number of pharmacist interventions/patient. The prescribing rates of antibiotics and their consumption levels were changed according to the NICU-specific antibiogram. There was a significant reduction in the 14-day and 28-day mortality of patients with late-onset sepsis after modifying the neonatal sepsis treatment protocol in the ASP intervention phase.

Conclusion:

ASP implementation was successful in improving antibiotic prescribing and patients outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Received antibiotics for more than 72 hours.

Exclusion Criteria:

* Hospital stay was less than 72 hours.
* Did not receive any antibiotics during hospital stay.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates admitted to NICU and received antibiotics for more than 72 hours
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
14-days mortality in each group | 6 months in the in the Pre-ASP phase and 6 months in the ASP intervention phase
  Number of patients who died from neonatal sepsis at the 14th day of their hospital stay was compared in the Pre-ASP phase and the ASP intervention phase
28-days mortality in each group | 6 months in the in the Pre-ASP phase and 6 months in the ASP intervention phase
  Number of patients who died from neonatal sepsis at the 28th day of their hospital stay was compared in the Pre-ASP phase and the ASP intervention phase

SECONDARY OUTCOMES:
Average Length of hospital stay in each group | 6 months in the in the Pre-ASP phase and 6 months in the ASP intervention phase
  In days
30-day readmission in each group | 6 months in the in the Pre-ASP phase and 6 months in the ASP intervention phase
  number of patients readmitted within 30 days from discharge

CONTACTS AND LOCATIONS:
Overall Officials: Neveen H. Abdelaal, M.sc., Principal Investigator — Department of Pharmacy and Medical Supplies, Assiut University Children's Hospital, Egypt; Nafisa H. Abdel Aziz, PhD, Study Chair — Department of Pediatrics, Faculty of Medicine, Assiut University, Egypt; Asmaa M. Abdelaziz, PhD, Study Chair — Department of Clinical Pathology, Faculty of Medicine, Assiut University, Egypt; Sahar B. Khalil, PhD, Study Director — Department of Clinical Pharmacy, Faculty of Pharmacy, Assiut University, Egypt; Mohamed M Abdel-Latif, PhD, Study Director — Department of Clinical Pharmacy, Faculty of Pharmacy, Assiut University, Egypt
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared